CLINICAL TRIAL: NCT01084551
Title: A Phase 3 Multi-Center, Placebo-Controlled, Double Blind, 3-Armed Parallel Group, Comparative Study of SPM 962 4.5 and 6.75 mg/Day to Investigate Superiority to Placebo in Patients With Restless Legs Syndrome
Brief Title: Study of SPM 962 in Patients With Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 243-09-001; JapicCTI-101053
Record Dates: First submitted 2010-03-04; First posted 2010-03-10 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-05

CONDITIONS: Idiopathic Restless Legs Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SPM 962 4.5 (Experimental): started at 2.25 mg/day to 4.5 mg/day for 13 weeks
  Interventions: Drug: SPM 962
- SPM 962 6.75 (Experimental): started at 2.25 mg/day to 6.75 mg/day for 13 weeks
  Interventions: Drug: SPM 962
- placebo (Placebo Comparator): for 13 weeks
  Interventions: Drug: Placebo of SPM 962

INTERVENTIONS:
Drug: SPM 962 — once a daily transdermal administration started at 2.25 mg/day to 4.5 mg/day for 13 weeks
  Arms: SPM 962 4.5
Drug: SPM 962 — once a daily transdermal administration started at 2.25 mg/day to 6.75 mg/day for 13 weeks
  Arms: SPM 962 6.75
Drug: Placebo of SPM 962 — once a daily transdermal administration for 13 weeks
  Arms: placebo

SUMMARY:
The objective of this study is to evaluate the clinical efficacy and safety of SPM962 in patients with restless legs syndrome (RLS) with once-daily repeated doses of 4.5mg and 6.75mg during a 13-week dose-titration and maintenance period. This is a multi-center, randomized, placebo-controlled, double-blind, 3-armed parallel group comparison study.

Efficacy will be determined by investigating the superiority of SPM962 to placebo in terms of the primary efficacy variable, change in International Restless Legs Syndrome Rating Scale (IRLS) total score from baseline to the end of the dose-maintenance period.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose condition has been diagnosed as RLS by meeting all 4 of the International Restless legs Syndrome Study Group/ National Institute of Health (IRLSSG/NIH) criteria
* Patients who meet any of the following criteria relating to RLS treatment:

  * Patients who have never received treatment for RLS
  * Patients who have received treatment for RLS in the past and responded to L-dopa or dopamine agonists (Response to other RLS medicines is irrelevant.)
* Patients who have an IRLS total score of >=15 at baseline
* Patients who experience symptoms in the evening or during the night on at least two days a week within 14 days prior to commencement of study treatment
* Patients and their partners can practice contraception at the end of follow-up observation period or by 1 week after the end of treatment

Exclusion Criteria:

* Patients who have previously participated in a clinical trial of SPM962 and taken the investigational product (IP)
* Patients with secondary RLS induced by renal impairment (uremia), iron deficiency anemia, drugs, pregnancy, etc.
* Patients who currently suffer, are at risk of developing, or have a history of sleep disorder such as sleep apnea syndrome, narcolepsy, and sleep attacks/sudden onset of sleep
* Patients who have concomitant diseases or symptoms which may affect the symptoms of RLS, such as polyneuropathy (including diabetic neuropathy), akathisia, claudication, varicoses, muscle fasciculation, painful legs and moving toes syndrome, radiculopathy and folate deficiency
* Patients who have other CNS diseases such as Parkinson's disease, dementia, progressive supranuclear paresis, multisystem atrophy, Huntington's Chorea, amyotrophic lateral sclerosis, and Alzheimer's disease
* Patients who have psychiatric conditions such as confusion, hallucination, delusion, and excitation, or patients who have abnormal behavior such as delirium, obsessive compulsive disorder, and impulse control disorder at the time of the screening test or baseline examination
* Patients whose SBP declines by at least 30 mmHg from supine to standing position based on the orthostatic hypotension assessment, or patients who develop orthostatic hypotension at baseline
* Patients who have a history of epilepsy, convulsion, etc
* Patients who have complications or a history of serious cardiac diseases or arrhythmia (eg, congestive heart failure of class 3 or 4 in the NYHA classification, second or third degree atrioventricular block, complete left bundle branch block, sick sinus syndrome, ventricular fibrillation, myocardial infarction within 12 months prior to the screening test, or a complication of angina pectoris)
* Patients with arrhythmia who have been taking Class 1a antiarrhythmic drugs (eg., quinidine, procainamide) or Class 3 antiarrhythmic drugs (eg., amiodarone, sotalol)
* Patients who have a serious ECG abnormality at the screening test and at the baseline examination

  * Patients who show QTc intervals exceeding 450 ms in both ECGs in the screening test
  * Patients who have an average QTc interval from the two ECGs in the baseline assessment that exceeds 470 ms (for females) or 450 ms (for males)
* Patients with congenital long QT syndrome
* Patients whose serum potassium level is < 3.5mEq/L at the screening test
* Patients whose total bilirubin is >= 3.0mg/dL, or whose AST(GOT) and ALT(GPT) are equal or more than 2.5 times the reference range of the clinical site (or >= 100IU/L) at the screening test
* Patients whose BUN level is >= 30mg/dL, or whose serum creatinine level is >= 2.0mg/dL at the screening test
* Patients who have a history of allergy to topical agents such as transdermal patch
* Patients who are pregnant or nursing or who wish to become pregnant during the study period
* Patients who habitually drink alcohol or smoke excessively
* Patients who engage in evening shift work or other such shift work, or whose work or circumstances makes it difficult to maintain a regular period of sleep
* Patients who engage in hazardous work such as driving a vehicle, operating machinery, or working in a high location.
* Patients with autoimmune disease, chronic active hepatitis, or immune deficiency disorder
* Patients who have a complication or history of malignant neoplastic disease, or received treatment for the disease within 12 months prior to the screening test
* Patients who are unable to properly record information in a patient diary
* Patients who received other IPs within 12 weeks prior to commencement of study treatment
* Patients who have been judged by the investigator or the sub-investigator to be inappropriate for inclusion in the study for any other reasons

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

REFERENCES:
- [Derived] Inoue Y, Shimizu T, Hirata K, Uchimura N, Ishigooka J, Oka Y, Ikeda J, Tomida T, Hattori N; Rotigotine Trial Group. Efficacy and safety of rotigotine in Japanese patients with restless legs syndrome: a phase 3, multicenter, randomized, placebo-controlled, double-blind, parallel-group study. Sleep Med. 2013 Nov;14(11):1085-91. doi: 10.1016/j.sleep.2013.07.007. Epub 2013 Aug 21. PMID 24055212

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 0 mg/day for 13 weeks
Period: Overall Study
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Started | 95 | 95 | 94
Completed | 86 | 81 | 86
Not Completed | 9 | 14 | 8
Not completed — Adverse Event | 2 | 9 | 4
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Protocol Violation | 2 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75 | Total
Number analyzed (Participants) | 95 | 95 | 94 | 284
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (15.3) | 50.7 (13.3) | 50.9 (13.7) | 51.7 (14.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 65 | 77 | 77 | 219
  >=65 years | 30 | 18 | 17 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 46 | 154
  Male | 41 | 41 | 48 | 130
Region of Enrollment [Number; unit: participants]
  Japan | 95 | 95 | 94 | 284

OUTCOME MEASURES:

1. Primary Outcome: International Restless Legs Syndrome Rating Scale (IRLS) Total Score
Description: Change from the baseline to the end of dose-titration/dose-maintenance period. IRLS is a scale for assessing severity of restless legs syndrome symptoms. IRLS consists of ten questions. Each question is scored from 4 for the first (top) answer (usually 'very severe') to 0 for the last answer (usually none).
  The sum of the score of each question serves as the scale score. The scale scoring criteria are: Mild (score 1-10); Moderate (score 11-20); Severe (score 21-30); Very severe (score 31-40). A decrease in the scores means improvement.
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (week 13)
Population: Full analysis set (FAS), last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Placebo: Once a daily transdermal administration for 13 weeks
- SPM 962 4.5: Once a daily transdermal administration of SPM 962 started at 2.25 mg/day to 4.5 mg/day for 13 weeks
- SPM 962 6.75: Once a daily transdermal administration of SPM 962 started at 2.25 mg/day to 6.75 mg/day for 13 weeks
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 95 | 93 | 94
Scores on a scale | -11.6 (8.2) | -14.3 (8.9) | -14.6 (9.0)

2. Secondary Outcome: Clinical Global Impression (CGI) Improvement
Description: CGI improvement is a clinician-reported scale for assessing how much the patient's illness has improved or worsened from baseline.
  The scale scoring criteria are 1: very much improved, 2: much improved, 3: minimally improved, 4: no change, 5: minimally worse, 6: much worse, 7: very much worse.
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (week 13)
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 95 | 93 | 93
Percentage of Participants
  Subjects with "much improved" | 24.2 | 25.8 | 29.0
  Subjects with "very much improved" | 33.7 | 41.9 | 45.2

3. Secondary Outcome: Patient Global Impression (PGI) Improvement
Description: PGI improvement is a patient-reported scale for assessing how much the patient's illness has improved or worsened from baseline.
  The scale scoring criteria are 1: very much better, 2: much better, 3: a little better, 4: no change, 5: a little worse, 6: much worse, 7: very much worse.
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (week 13)
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 95 | 93 | 93
Percentage of Participants
  Subjects with "much improved" | 23.2 | 24.7 | 30.1
  Subjects with "very much improved" | 38.9 | 48.4 | 50.5

4. Secondary Outcome: The Pittsburgh Sleep Quality Index (PSQI)
Description: Change of PSQI from baseline to the end of dose-titration/dose-maintenance period.
  PSQI is a scale for assessing severity of sleep disorders. The score ranges from 0 to 21. 0 indicates "no difficulty" and 21 indicates "severe difficulty". A decrease in the scores means improvement.
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (week 13)
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 94 | 93 | 90
Scores on a scale | -2.5 (2.4) | -3.1 (3.2) | -3.2 (3.3)

5. Secondary Outcome: Each Item of IRLS (10 Items)
Description: IRLS is a scale for assessing severity of restless legs syndrome symptoms. IRLS consists of ten questions. Each question is scored from 4 for the first (top) answer (usually 'very severe') to 0 for the last answer (usually none).
  Numbers of subjects with -4 or -3 score change from baseline in each item of IRLS. A decrease in the scores means improvement.
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (week 13)
Population: FAS, LOCF
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 95 | 93 | 94
percentage of participants
  -4 (RLS discomfort) | 1.1 | 2.2 | 6.4
  -3 (RLS discomfort) | 11.6 | 17.2 | 12.8
  -4 (need to move around due to RLS symptoms) | 2.1 | 2.2 | 7.4
  -3 (need to move around due to RLS symptoms) | 11.6 | 25.8 | 18.1
  -4 (discomfort relief by moving around) | 0 | 1.1 | 2.1
  -3 (discomfort relief by moving around) | 10.5 | 20.4 | 28.7
  -4 (severity of RLS as a whole) | 1.1 | 1.1 | 4.3
  -3 (severity of RLS as a whole) | 6.3 | 12.9 | 12.8
  -4 (RLS symptoms frequency) | 12.6 | 24.7 | 26.6
  -3 (RLS symptoms frequency) | 12.6 | 9.7 | 11.7
  -4 (average duration of RLS symptoms) | 1.1 | 2.2 | 2.1
  -3 (average duration of RLS symptoms) | 6.3 | 10.8 | 9.6
  -4 (severity of sleep disturbance) | 2.1 | 4.3 | 6.4
  -3 (severity of sleep disturbance) | 16.8 | 16.1 | 21.3
  -4 (tiredness or sleepiness during the day) | 0 | 2.2 | 2.1
  -3 (tiredness or sleepiness during the day) | 8.4 | 11.8 | 8.5
  -4 (severity of the impact on daily affairs) | 0 | 1.1 | 1.1
  -3 (severity of the impact on daily affairs) | 8.4 | 11.8 | 4.3
  -4 (severity of mood disturbance) | 1.1 | 4.3 | 1.1
  -3 (severity of mood disturbance) | 8.4 | 10.8 | 12.8

6. Secondary Outcome: Incidence of RLS Symptoms
Description: Incidence rate of RLS symptoms is calculated as the number of days with RLS symptoms in the week / the number of evaluation days in the week* 100%
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (week 13)
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: percentage of days with RLS symptom
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 95 | 93 | 92
percentage of days with RLS symptom
  Baseline | 85.7 (20.8) | 85.4 (20.5) | 83.2 (22.2)
  Week 13 | 48.7 (40.9) | 35.8 (38.6) | 36.8 (38.8)

7. Secondary Outcome: Average Duration of RLS Symptoms
Description: Change of average duration of RLS symptoms in a week from baseline to the end of dose-titration/dose-maintenance period. Only the days with RLS symptoms are used for calculation.
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (weeks 13)
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 71 | 59 | 55
Hours | -3.1 (4.7) | -3.7 (4.6) | -4.3 (4.4)

8. Secondary Outcome: Incidence of RLS Symptoms in the Evening and Night
Description: Incidence rate of RLS symptoms is calculated as the number of days with RLS symptoms / the number of days of evaluation * 100%.
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (week 13)
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: percentage of days/week with symptoms
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 95 | 93 | 92
percentage of days/week with symptoms
  Baseline | 80.6 (24.2) | 83.3 (20.8) | 79.5 (24.2)
  Week 13 | 45.4 (41.0) | 34.6 (38.2) | 31.8 (37.7)

9. Secondary Outcome: Average Duration of RLS Symptoms in the Evening and Night in a Week
Description: as for outcome 7
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (weeks 13)
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 69 | 58 | 50
Hours | -1.3 (3.1) | -1.8 (2.5) | -1.5 (2.3)

10. Secondary Outcome: Nocturnal Awakenings Due to RLS Symptoms in a Week
Description: Nocturnal awakening rate is calculated as the number of days with nocturnal awakenings / the number of days of evaluation * 100%.
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (week 13)
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: percentage of days/week with awakening
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 95 | 93 | 92
percentage of days/week with awakening
  Baseline | 33.5 (35.9) | 22.6 (31.3) | 28.3 (34.3)
  Week 13 | 15.6 (31.7) | 7.7 (20.5) | 7.5 (19.5)

11. Secondary Outcome: Average Sleep Time in a Week
Description: Change of average sleep time in a week from baseline to the end of dose-titration/dose-maintenance period.
Time Frame: Baseline, the end of dose-titration/dose-maintenance period (weeks 13)
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Number analyzed (Participants) | 95 | 93 | 92
Hours | 0.4 (0.8) | 0.5 (1.1) | 0.4 (1.1)

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Placebo | SPM 962 4.5 | SPM 962 6.75
Serious Adverse Events (participants affected / at risk) | 2/95 | 0/95 | 1/94
Other Adverse Events (participants affected / at risk) | 32/95 | 72/95 | 77/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=95) | SPM 962 4.5 (N=95) | SPM 962 6.75 (N=94)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lacunar Infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
VIIth Nerve Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=95) | SPM 962 4.5 (N=95) | SPM 962 6.75 (N=94)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 9 (12) | 32 (37) | 41 (48)
Vomiting (Gastrointestinal disorders) | 1 (2) | 4 (5) | 10 (11)
Abdominal Discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0) | 10 (11)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Application Site Reaction (General disorders) | 7 (8) | 40 (41) | 47 (50)
Malaise (General disorders) | 1 (2) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 12 (17) | 12 (14) | 16 (17)
Headache (Nervous system disorders) | 0 (0) | 5 (6) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Somnolence (Psychiatric disorders) | 2 (2) | 10 (10) | 14 (14)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No